CLINICAL TRIAL: NCT00279162
Title: Calcipotriene Plus Betamethasone Dipropionate Gel Compared to the Gel Vehicle in Scalp Psoriasis, in Patients Receiving Calcipotriene Plus Betamethasone Dipropionate Ointment for Psoriasis Vulgaris of Trunk/Limbs
Brief Title: Efficacy and Safety of Calcipotriene/Betamethasone Gel/Ointment in Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MBL 0502 US
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2015-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — calcipotriene; Ointments

INTERVENTIONS:
Drug: Calcipotriene/betamethasone gel and ointment

SUMMARY:
Patients will receive either a gel containing both calcipotriene plus betamethasone or gel with no active ingredients as treatment for their scalp psoriasis for 8 weeks. After this time all patients will receive the gel containing both calcipotriene and betamethasone for 44 weeks. In addition, patients will receive an ointment containing both calcipotriene plus betamethasone as treatment for their psoriasis of the trunk and limbs for 52 weeks.

The objective is to study the short-term efficacy of the gel, and the short and long-term safety of the gel and the ointment.

ELIGIBILITY:
Inclusion Criteria:

* Psoriasis involving at least 10% of the scalp and amenable to topical treatment with a maximum of 40g of gel per week.
* A score for the investigator's assessment of clinical signs of scalp psoriasis of at least 2 (moderate severity) in one of the clinical signs (redness, thickness and scaliness), and at least 1 (slight severity) in each of the other two clinical signs.
* An investigator's global assessment of moderate, severe or very severe scalp psoriasis.
* Psoriasis vulgaris of the trunk and/or limbs amenable to topical treatment with a maxi-mum of 60g of ointment per week.
* An investigator's global assessment of moderate, severe or very severe psoriasis of trunk/limbs.
* Attending a hospital out-patient clinic or the private practice of a dermatologist for treatment of psoriasis.
* Patients who self-report: - their ethnicity as Hispanic or Latino, and who are of any race, - their ethnicity as not Hispanic or Latino, and their race as Black or African American.
* Following receipt of verbal and written information about the trial, the patient must provide signed and dated informed consent before any trial-related activity is carried out.
* Females of child-bearing potential must have a negative result for a urine pregnancy test before randomisation and must agree to use an adequate method of contraception during the study.
* Patients fulfilling US requirements/law for participation in this study.

Exclusion Criteria:

* PUVA or Grenz ray therapy within 4 weeks prior to randomisation.
* UVB therapy within 2 weeks prior to randomisation.
* Systemic treatment with biological therapies (marketed or otherwise) with a possible effect on psoriasis (e.g., alefacept, efalizumab, etanercept, infliximab) within 3 months prior to randomisation.
* Systemic treatment other than biologicals with a possible effect on psoriasis (e.g., corticosteroids, vitamin D analogues, retinoids, hydroxycarbamide, azathioprine, meth-otrexate, cyclosporine, other immunosuppressants) within 4 weeks prior to randomisation.
* Any topical treatment of the scalp (except for medicated shampoos and emollients) within 2 weeks prior to randomisation (medicated shampoos/emollients are not allowed during the double-blind phase). Shampoos containing corticosteroids, e.g. Clobex®, are not allowed within 2 weeks prior to randomisation.
* Planned use of topical treatment for psoriasis of the trunk or limbs, besides study medication, during the study with the exceptions of: • emollient • medications used to treat psoriasis of the skin folds and/or genitals (any medication may be used for this purpose apart from Class 1-5 corticosteroids.
* Topical treatment of the face with Class 1-5 corticosteroids within 2 weeks prior to randomisation.
* Planned initiation of, or changes to, concomitant medication that could affect psoriasis (e.g., beta blockers, anti-malaria drugs, lithium) during the double-blind phase of the study.
* Treatment with any non-marketed drug substance (i.e., an agent which has not yet been made available for clinical use following registration) within 4 weeks prior to randomisation.
* Planned use of chemical treatments of the hair (eg relaxers, 'perms', or colourings) during the double-blind phase of the study.
* Current diagnosis of erythrodermic, exfoliative or pustular psoriasis.
* Patients with any of the following conditions also present on psoriatic areas of the scalp or trunk/limbs: viral (e.g. herpes or varicella) lesions of the skin, fungal or bacterial skin infections, parasitic infections, skin manifestations in relation to tuberculosis or syphilis, rosacea, acne rosacea, acne vulgaris, atrophic skin, striae atrophicae, fragility of skin veins, ichthyosis, ulcers or wounds.
* Other inflammatory skin diseases that may confound the evaluation of psoriasis of the scalp or trunk/limbs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2005-12; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy (in terms of patients with clear or minimal disease) of 8 weeks treatment with combination (calcipotriene plus betamethasone dipropionate) gel with that of the gel vehicle in scalp psoriasis.

SECONDARY OUTCOMES:
To compare the safety of 8 weeks treatment with combination gel with that of the gel vehicle in scalp psoriasis.
To evaluate the efficacy and safety of 4 weeks treatment with combination ointment in psoriasis vulgaris of trunk/limbs.
To evaluate the safety of 52 weeks treatment (used when required) with combination gel in scalp psoriasis.
To evaluate the safety of 52 weeks treatment (used when required) with combination ointment in psoriasis vulgaris of trunk/limbs.

CONTACTS AND LOCATIONS:
Overall Officials: S Tyring, MD, Principal Investigator — Center for Clinical Studies
Locations (1):
- Center for Clinical Studies, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en